CLINICAL TRIAL: NCT02766699
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, and Immunogenicity of EGFR (Vectibix® Sequence)-Targeted EnGeneIC Dream Vectors Containing Doxorubicin (EGFR(V)-EDV-Dox) in Subjects With Recurrent Glioblastoma Multiforme (GBM)
Brief Title: A Study to Evaluate the Safety, Tolerability and Immunogenicity of EGFR(V)-EDV-Dox in Subjects With Recurrent GBM
Acronym: CerebralEDV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Engeneic Pty Limited (Industry)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENG7
Record Dates: First submitted 2016-05-03; First posted 2016-05-10 (Estimated); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Glioblastoma; Astrocytoma, Grade IV
Keywords: Astrocytoma, Grade IV; Doxorubicin; Glioblastoma; Neoplasms; Neoplasms by Site; Antineoplastic Agents; Drug Delivery Systems; Molecular Targeted Therapy; Nanoparticles; Disease Progression; Recurrence; Brain Neoplasms; Immunotherapy; Receptor, Epidermal Growth Factor; Antibodies, Bispecific
MeSH Terms: conditions — Glioblastoma; Neoplasms; Neoplasms by Site; Disease Progression; Recurrence; Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: 3+3 dose escalation study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- EGFR(V)-EDV-Dox (Experimental): EGFR(V)-EDV-Dox administered via 20 minute intravenous infusion once a week for seven weeks (1 Cycle). Subjects will receive one of two dose levels: 5 x 10^9 or 8 x 10^9. All subjects will undergo an adapted dose escalation regime in the first cycle of treatment. For subsequent cycles all doses will be administered at full strength (5x10^9 or 8x10^9 EGFR(V)-EDV-Dox). Subjects may receive further cycles of treatment if the tumor remains stable or is responding, and/or they are deriving clinical benefit from the therapy and are tolerating treatment.
  Interventions: Drug: EGFR(V)-EDV-Dox

INTERVENTIONS:
Drug: EGFR(V)-EDV-Dox — EGFR(V)-EDV-Dox using EnGeneIC EDV™ technology is a bacterially derived minicell which packages a toxic payload, Doxorubicin, into a 400 nm particle which targets specific cancer cells using bispecific antibodies (BsAb). BsAb-targeted, payload-packaged EDV nanocells only exit the leaky blood vessels associated with tumors and enter into the tumor microenvironment. The BsAb binds to the tumor cell-surface receptor, where the EDV is taken up, broken down within the cancer cell and releases the Doxorubicin. The residual EDVs that do not make it into the tumor microenvironment, are engulfed by cells of the immune system and since the EDVs are derived from bacteria, they carry potent immuno-stimulating components which appear to bypass the immuno-suppression caused by the tumor.
  Other Names: EnGeneIC Dream Vector™; EnGeneIC Delivery Vehicle™

SUMMARY:
The purpose of the Cerebral EDV study is to determine the safety and tolerability of EGFR(V)-EDV-Dox in order to establish the best dose level to be used in future studies. The study will also examine the body's immune response to EGFR(V)-EDV-Dox and assess if it is effective in the treatment of patients with recurrent glioblastoma multiforme (GBM).

DETAILED DESCRIPTION:
This is an open-label, Phase 1, dose exploration and preliminary immunogenicity study of single agent EGFR(V)-EDV-Dox in subjects with recurrent glioblastoma (GBM). Eligible subjects enrolled in the study will receive EGFR(V)-EDV-Dox administered weekly for 7 weeks via IV 20 minute infusion, followed by radiological evaluation at week 8 (1 Cycle). Subjects may continue to receive subsequent cycles of EGFR(V)-EDV-Dox unless the subject becomes intolerant to investigational product (IP), withdraw consent or the individual is no longer receiving clinical benefit (factors taken in to consideration will be disease progression radiologically or clinically, and clinical benefits to quality of life). Tumour assessment will be repeated after each 7 week cycle (week 8).

The study will take place in two parts, Part 1 (Dose Exploration) and Part 2 (Dose Expansion).

Part 1 - Dose Exploration will assess the safety and tolerability of multiple doses of drug at two dose levels (5 x 10^9 and 8 x 10^9) and will enroll prior to Part 2. Three subjects will be recruited per dose level. Enrollment will begin with the 5 x 10^9 dose level, and the decision to enroll to the 8 x 10^9 dose level will follow a comprehensive safety evaluation and a standard 3 + 3 dose escalation study design.

Part 2 - Dose Expansion will be conducted pending safety results of Part 1 to provide guidance regarding the recommended phase 2 dose (RP2D). Subjects will be treated and assessed as outlined in Part 1 above. If 0 out of 3 subjects, or 1 out of 6 subjects, experience dose limiting toxicities (DLTs) at the 5 x 10^9 dose level in Part 1, additional subjects to a total of 10 will be recruited to this dose level in Part 2. Similarly, if 0 out of 3 subjects, or 1 out of 6 subjects, experience DLTs at the 8 x 10^9 dose level in Part 1, additional subjects to a total of 10 will be recruited to this dose level in Part 2. If both dose levels are tolerated, a total of 10 subjects per dose level will be enrolled.

A safety follow-up visit must be performed 30 (+5) days after the last dose of drug for all subjects.All subjects who discontinue investigational product and who have not withdrawn full consent to participate in the study will continue in the long term follow-up phase. Long term follow-up will continue approximately every 1 month for 12 months, from the 30 (+5) day follow-up visit, then approximately every 2-3 months for the extent of subject survival.

ELIGIBILITY:
Inclusion Criteria:

1. Karnofsky Performance Status (KPS) ≥ 60%.
2. Life expectancy ≥ 3 months.
3. Pathologically documented, and definitively diagnosed recurrent World Health Organization (WHO) Grade IV astrocytoma (GBM).
4. Participant must have archived tumor tissue available from initial diagnosis or subsequent relapse(s) of Grade IV GBM for submission for central review at Investigational sites local laboratories.
5. Recurrence or progression of disease (confirmed by MRI and measurable by RANO criteria) following receipt of standard of care therapy, which includes maximum safe surgical resection, standard adjuvant radiation/temozolomide treatment. Participants must have completed at least 21 days of temozolomide treatment in combination with radiation therapy to be considered to have received standard of care therapy.
6. Participant has received no more than 1 other therapeutic regimen other than those listed above in (5).
7. Participant may be receiving steroid therapy at time of enrollment (stable dose of ≤ 4 mg/day of dexamethasone or steroid equivalent).
8. Ability to undergo MRI evaluation.
9. Participant has ≥ 1 site of bi-dimensionally measurable disease measured using contrast enhanced MRI.
10. Hematological function:

    * White blood cell count (WBC) ≥ 3.0 x 109/L
    * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
    * Platelet count ≥ 100 x 109/L
    * Hemoglobin > 9 g/dL
    * Prothrombin time (PT) or partial thromboplastin time (PTT) < 1.5 x upper limit of normal (ULN)
    * International normalized ratio (INR) < 1.5 x ULN
11. Renal function:

    * Blood urea nitrogen (BUN) < 30 mg/dL
    * Creatinine serum levels ≤ 1.5 x ULN
    * Or creatinine clearance ≥ 60 mL/minute for subjects with serum creatinine outside the normal range (calculated using the Cockcroft-Gault equation).
12. Hepatic function:

    * Aspartate aminotransferase (AST) < 2.5 x ULN (3 x ULN for subjects on chronic anticonvulsive therapies known to increase transaminases).
    * Alanine aminotransferase (ALT) < 2.5 x ULN (3 x ULN for subjects on chronic anticonvulsive therapies known to increase transaminases).
    * Alkaline phosphatase (ALP) < 2.5 x ULN (3 x ULN for subjects on chronic anticonvulsive therapies).
    * Total bilirubin ≤ 1 x ULN (unless elevated due to Gilbert's syndrome or extrahepatic source as denoted by increased indirect bilirubin fraction. Subjects with ≥1 x ULN will be tested for direct bilirubin fraction so that the indirect fraction can be calculated).
13. Adequate cardiac function with left ventricular ejection fraction (LVEF) ≥ 55% at baseline.
14. Serum phosphate levels that are within normal limits (2.4 - 4.1 milligrams per deciliter mg/dL) at baseline.
15. Subject meets the reproductive criteria as follows:

    * Female subjects who are of non-reproductive potential (ie, post menopausal by history - no menses for ≥ 1 year and follicle-stimulating hormone (FSH) level consistent with post-menopausal status; OR history of hysterectomy; OR history of bilateral tubal ligation; OR history of bilateral oophorectomy).
    * Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days prior to the 1st dose, if more than 7 days prior, a urine pregnancy test must be performed before the 1st dose. The female subject must be willing to use highly effective methods of birth control during the period of therapy and for 6 months following the last study IP administration. Highly effective methods of birth control include sexual abstinence, hormonal birth control, or intrauterine device (women), vasectomy or a condom with spermicide (men) in combination with barrier methods.
    * Male subjects who are willing to use highly effective methods of birth control during the period of therapy and for 6 months following the last IP administration.
    * All study subjects must be willing to ensure that corresponding sexual partners practice these same methods of highly effective birth control for the same duration.

Exclusion Criteria:

1. History of central nervous system bleeding as defined by stroke or intraocular bleed within 6 months of enrollment.
2. Evidence of acute intracranial / intra-tumoral hemorrhage, except for participants with stable grade 1 hemorrhage.
3. History of coronary artery disease, with or without angina pectoris or myocardial infarction, symptomatic congestive heart failure (New York Heart Association > Class II), uncontrolled hypertension (systolic > 160 mmHg or diastolic > 100 mmHg) or cardiac arrhythmias requiring anti-arrrhythmic therapy.
4. Clinically significant electrocardiogram (ECG) changes at enrollment which obscure the ability to assess the PR, QT, and QRS interval; congenital long QT syndrome.
5. Active infection requiring treatment.
6. History of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer, or other malignancies curatively treated with no evidence of disease for ≥ 2 years.
7. Known positive test for human immunodeficiency virus infection (HIV), or active hepatitis B or hepatitis C infection.
8. Receipt of therapies or procedures prior to first dose including:

   * Radiation therapy within 6 months of Study Day 1 or has not recovered from the toxic effects of such therapy.
   * Bevacizumab® or other anti-angiogenic therapy.
   * Gliadel® Wafer (within 6 months of Study Day 1, or has not recovered from the toxic effects of such therapy).
   * Immunotherapeutic agents, vaccines, or monoclonal antibody therapy (within 4 weeks of Study Day 1 or has not recovered from the toxic effects of such cancer therapy).
   * Temozolomide or other chemotherapy (within 4 weeks of Study Day 1 or 6 weeks for nitrogen mustards, or has not recovered from the toxic effects of such cancer therapy).
   * Anticoagulation therapy (within 7 days of Study Day 1), except low molecular weight heparins or low dose aspirin.
   * Other investigational therapy (within 30 days of Study Day 1).
   * Surgical resection of brain tumor (within 4 weeks of Study Day 1 or has not recovered from acute side effects of such therapy except for neurological effects).
   * Any major surgery (within 4 weeks of Study Day 1, or has not recovered from the effects of such surgery).
9. Subject has a known allergic/hypersensitivity to investigational components or excipients (doxorubicin, trehalose, monoclonal antibody therapy, penicillin class of antibiotics, gentamicin (or other aminoglycosides), or ciprofloxacin hydrochloride (or other quinolones)).
10. If female, is pregnant or is breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-10-25 (Actual); Primary Completion 2021-08-21 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Safety outcome measures | Safety measures will be conducted from Study Day 1 as per study schedule to safety follow-up visit 30 (+5 days) post last dose.
  Recording of adverse Events (AE's) and clinically significant changes in vital signs, physical and neurological examinations, cardiac tests, radiological imaging inc. CT scan (Day 27/28) and clinical laboratory tests.

SECONDARY OUTCOMES:
Efficacy outcome measure | Screening, then post cycle (Days 50-56)
  Disease response will be measured by Magnetic Resonance Imaging (MRI) using Response Assessment in Neuro-Oncology (RANO).
Identification of a recommended Phase 2 dose (RP2D) of EGFR(V)-EDV-Dox in subjects with recurrent GBM | DLT evaluable subjects are those who experience a DLT assessed within the first treatment cycle of Part 1 i.e.including up to 7 days after the final dose, days 1-50 of treatment.
  Review of safety data for dose limiting toxicity (DLT) evaluable subjects.
Overall survival outcome measure | The number of days from the date of first administration of EGFR(V)-EDV-Dox to the date of death, regardless of cause up to 60 months.
  Overall survival is defined as time from the date of first administration of EGFR(V)-EDV-Dox to the date of death, regardless of cause

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer MacDiarmid, Ph.D, Study Director — Engeneic Pty Limited; Himanshu Brahmbhatt, Ph. D, Study Director — Engeneic Pty Limited; Gary L Gallia, M.D., Ph.D, Principal Investigator — Johns Hopkins University; Stuart A Grossman, M.D., Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - John Hopkins Hospital, Baltimore, Maryland
  - Lenox Hill Hospital, Northwell Health, New York, New York

IPD SHARING:
Plan to Share IPD: No